CLINICAL TRIAL: NCT04307108
Title: Evaluation of the Acceptability and Usability of the MAGIC-GLASS Solution as Part of the Care Pathway in People With Acute, Sub-Acute and Chronic Stroke
Brief Title: Magic Glass Evaluation in People With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Western Health and Social Care Trust (Other); Southern Health and Social Care Trust (Other Government); Tech 4 Care (Unknown); miThings AB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/NI/0080
Record Dates: First submitted 2020-02-17; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: stroke, virtual reality, upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magic Glass — MAGIC-GLASS is a VR-based home system for stroke rehabilitation, developed by Ulster University (UK) in collaboration with Tech4Care srl (Italy) and miThings AB (Sweden) in the context of the EU-funded Project Magic (grant agreement No 687228). It includes a number of mini-games grounded on rehabilitation paradigms such as mirror therapy [29] and can adapt to the capability of a person. In addition, the games will include an automatic coaching system for giving feedback both on rehabilitation results (e.g. achievement of exercise goals) and performance (during the exercise itself, the system will give real time advice on the execution of the exercise).

SUMMARY:
Background: Virtual Reality (VR) technology may help to provide a way for stroke survivors to exercise in their own time at home, with remote clinical support. Before we introduce this technology we need to test that it will work alongside current health services for stroke survivors. Aims: To find out if using the MAGIC-GLASS solution alongside current healthcare care is usable and acceptable to stroke survivors and helps to increase rehabilitation time. Design: Measures before and after stroke survivors use the MAGIC-GLASS solution.

Setting: Stroke survivors will use the MAGIC-GLASS solution in their own home. Population: adults (≥18 years) who have had a stroke at least two weeks before they enter into the study.

Interventions: Our VR technology is called MAGIC-GLASS, and in order to use the solution the user puts on a headset which is connected to a computer. They can then see a VR environment in which they will be able to see virtual hands that respond to the movements of their own hands. It will also be possible to see a mirror image of their hands moving. The system will record how much they use the system and improvement in their movement. Regular contact will be made with a clinician who will be able to use the system to see (from their clinic) how the stroke survivor is doing and talk to them. Outcomes: We want to find out how the stroke survivors' movement changes over time and what they think of using the system. We will also ask clinical staff what they thought of using the system as part of healthcare provision to stroke survivors. Finally we want to find out how much it will cost to use the system.

ELIGIBILITY:
Inclusion Criteria:

* Any time point post stroke
* Medically stable (and without uncontrolled seizures or vertigo)
* No or mild cognitive deficit: can follow two step commands
* No significant visual or spatial neglect (Can turn head towards an image when asked to do so and keep attention). People with hemianopia or other visual deficits can be included dependent on clinical opinion
* Normal or normal corrected vision
* Be able to get in and out from a seat with assistance; can be used in a wheelchair as long as arms can rest on table
* Have a carer to assist putting on the headset
* Be willing to give consent
* For those not using mirror therapy, can move impaired arm without significant pain

Exclusion Criteria:

* • People with a moderate to severe cognitive impairment (MoCA<20).

  * Those with a visual impairment who are unable to see a clear image with the headset.
  * Patients with severe neuropsychological deficits such as severe neglect or apraxia as indicated by their clinical team.
  * Patients who are medically unwell e.g. with history of solid organ or bone marrow transplantation, active malignancy within 24 months prior to screening or metastatic cancer, life expectancy less than 6 months, Congestive heart failure in New York Heart Association (NYHA) Functional Classification IV (severe) stage.
  * Those with complete dependency in Activities of Daily Living, any medical or other reason (e.g. known or suspected inability of the participant to comply with the protocol procedure) that investigator opinion that the participant is unsuitable for the study.
  * Patients unwilling to provide consent and those who cannot be followed-up at any time point will be excluded from the study.
  * Epilepsy, seizures and history of vertigo (possible exclusion determined by clinician).
  * Those with upper limb sensory disturbance who are unwilling to keep their nails short for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
the usability of the intervention; | through study completion, an average of 6 months
  Combination of interviews with users, carer questionnaire, focus groups with clinicians will be used to assess usability using qualitative analysis
the usability of the intervention | through study completion, an average of 6 months
  System usability score questionnaire
the acceptability of the intervention | through study completion, an average of 6 months
  Combination of interviews with users, carer questionnaire, focus groups with clinicians will be used to assess acceptability by analysing qualitatively
the process requirements for the new care pathway; | through study completion, an average of 6 months
  Combination of interviews with users, carer questionnaire, focus groups with clinicians and will be analysed qualitatively
the resource requirements for the new care pathway; | through study completion, an average of 6 months
  Combination of interviews with users, carer questionnaire, focus groups with clinician and will be analysed qualitatively
the intensity in Rehabilitation Therapy | Change from baseline to end of intervention (6 months)
  measured in clinical dashboard
the duration in Rehabilitation Therapy | Change from baseline to end of intervention (6 months)
  measured in clinical dashboard

SECONDARY OUTCOMES:
Functional independence in the activities of daily living with respect to the modified Rankin Scale | Change from baseline to end of intervention (6 months)
Functional independence in the activities of daily living with respect to the Barthel Index | Change from baseline to end of intervention (6 months)
physical activity as measured by range of motion | Change from baseline to end of intervention (6 months)
  measured by sensors inbuilt in the computer system
cognitive function | Change from baseline to end of intervention (6 months)
  Montreal Cognitive Assessment
Stroke specific quality of life | Change from baseline to end of intervention (6 months)
  Stroke specific quality of life questionnaire
potential cost effectiveness of the solution | Change from baseline to end of intervention (6 months)
  health care resource questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- Neuro-rehabilitation Department of the University Hospital of Ancona., Ancona, Italy
- United Kingdom (2):
  - Western Health and Social Care Trust, Londonderry
  - Southern Health and Social Care Trust, Lurgan

IPD SHARING:
Plan to Share IPD: No